CLINICAL TRIAL: NCT06352957
Title: Use of ETElcalcetidefor pReserving vitamiN K-dependent proteIn activiTY ITAlian Study
Acronym: ETERNITY-ITA
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Sponsor
Other Study IDs: 23022022CERC
Record Dates: First submitted 2024-03-21; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Matrix Gla protein; Osteocalcin or Bone GLA Protein (BGP); Vascular calcification; Vitamin K; Etecalcetide; Bone Fractures
MeSH Terms: conditions — Vascular Calcification; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Etecalcetide Group: Drug: Etelcalcetide Administered intravenously at the end of each dialysis session. Dosing ranges from 2.5 mg to 15 mg set by the patient's physician.
  Other Name: Parsabiv
- Standard of Care: Drug: Vitamin D or Vitamin D analogs

SUMMARY:
The goal of this Prospective Observational Study of comparative effectiveness is to provide real world evidence of the effect of Etelcalcetide in increasing actives form VKDPs levels such as BGP and MGP at 3, 9 and 18 months from baseline, with resulting correct bone mineralization and inhibition vascular calcification in hemodialysis patients.

The study will enroll 160 hemodialysis patients: 80 patients treated with Etelcalcetide and 80 age and sex matched patients treated with Calcitriol or vitamin D analogs. The treating nephrologist will base the target dose of Etelcalcetide on individual-level in order to achieve the KDIGO PTH target. In the Etelcalcetide-treated group, the addition of calcitriol will be allowed when required by clinical practice (for correction of hypocalcemia). The main endpoint is the comparison of the levels of active forms of VKDP (MGP and BGP) between patients treated with Etelcalcetide and those treated with vitamin D or vitamin D analogues. The measurements of the biomarkers are scheduled at baseline and after 3, 9, and 18 months.

DETAILED DESCRIPTION:
Vascular calcifications (VCs) are frequent complications of chronic kidney disease (CKD), and mineral disorders are associated with aortic calcifications and increased risk of bone fractures. The complex pathogenesis of VCs involves various factors such as calcium overload, phosphate imbalance, and secondary hyperparathyroidism. Key inhibitors, such as vitamin K-dependent proteins (VKDPs) like matrix Gla protein (MGP) play pivotal roles in VCs development. Traditional treatments to reduce VC focus on lowering PTH, calcium and phosphorus levels and etelcalcetide revealed as a promising therapy to this scope. Accordingly, the VItamin K Italian study (VIKI) reported that calcimimetics treated hemodialysis patients had higher levels of total BGP and MGP versus those untreated, suggesting a protective effect of this drugs class. These findings point out the multifactorial nature of VC in CKD and suggest new treatment strategies and targeted pathways for improving outcomes. The ETERNITY-ITA study will investigate the real world effect of Etelcalcetide in increasing actives form VKDPs levels such as BGP and MGP thus contributing to bone and vascular health in hemodialysis patients. ETERNITY-ITA is a multi-center comparative effectiveness, observational, longitudinal study. The study will enroll 160 hemodialysis patients: 80 patients treated with Etelcalcetide and 80 age and sex matched patients treated with Calcitriol or vitamin D analogs. The treating nephrologist will base the target dose of Etelcalcetide on individual-level in order to achieve the KDIGO PTH target. In the Etelcalcetide-treated group, the addition of calcitriol will be allowed when required by clinical practice (for correction of hypocalcemia). The main endpoint is the comparison of the levels of active forms of VKDP (MGP and BGP) between patients treated with Etelcalcetide and those treated with vitamin D or vitamin D analogues. The measurements of the biomarkers are scheduled at baseline and after 3, 9, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided informed consent;
2. Patient is 18 years of age or older of both gender;
3. Patients receiving maintenance HD three times per week (Kt/V >1.2);
4. Parathyroid hormone concentrations >500 ng/l at screening, or if parathyroidectomy is planned or expected, Ca >8.3 mg/dl;
5. Will be considered patients in the exposed group:

   1. Patients who have started Etelcalcetide within 1-month before the study enrolment;
   2. Patients naïve to intravenous calcimimetics use;
   3. Patients who have suspended oral calcimimetics from at least 1-month;
   4. Patients who are not responder or not compliant to the treatment with calcitriol;
6. In the unexposed group, patients on treatment with calcitriol or vitamin D analogs and who are age (± 2 years) and sex comparable (matching) to those in the exposed group will be considered;
7. Native vitamin D can be used in both groups and should be administered to target a 25(OH)D level > 30 ng/ml;
8. Dialysate calcium concentration must be stable for at least 4 weeks prior to screening laboratory assessments;
9. Patient must have severe HPT as defined by two laboratory screening pre-dialysis serum PTH values > 500 pg/ml, measured on two consecutive lab checks prior to entering the study. PTH levels should be standardized according to the following table (Souberbielle et al. Kidney Int 2010);
10. Total alkaline phosphatase greater than the normal range, or even within the normal range but if greater than the tertile of the reference range for the assay;
11. Patients will be eligible only if they will show at least a moderate Aorta VCs and/or Iliac arteries VCs and at least a mild VF.

Exclusion Criteria:

1. Previous treatment with oral calcimimetics (cinacalcet) must have been suspended for at least 30 days. Recent start of calcimimetics (Etelcalcetide) is acceptable, but patients are excluded if treatment lasts for more than 1 month;
2. Patients has received a bisphosphonate, denosumab or teriparatide during the 12 months prior to screening;
3. The patient underwent parathyroidectomy in the 6 months before the start of the study or if scheduled soon;
4. Scheduled kidney transplant during the study period or anticipated living donor evaluation within three months of recruitment;
5. Patient has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator;
6. Metabolic bone diseases not related to the kidney (i.e., Pagets, Osteogenesis Imprefecta);
7. Severe untreated hyperthyroidism;
8. Malignancy within the last 3 years (except non-melanoma skin cancers or cervical carcinoma in situ);
9. Patient is pregnant or nursing;
10. Patients with Long QT Syndrome;
11. Patient likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the patient and Investigator's knowledge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of VKDP | Baseline and after 3, 9, and 18 months of treatment
  The primary endpoint is the comparison of the levels of active forms of VKDP between patients treated with Etelcalcetide and those treated with vitamin D or vitamin D analogues (MGP and BGP).

SECONDARY OUTCOMES:
Calcium | Baseline, 3, 9 and 18-months
  Concentration of calcium (mg/dL)
Phosphate | Baseline, 3, 9 and 18-months
  Concentration of phosphate (mg/dL)
Magnesium | Baseline, 3, 9 and 18-months
  Concentration of magnesium (mg/dL)
ALP | Baseline, 3, 9 and 18-months
  Concentration of ALP (U/L)
PTH | Baseline, 3, 9 and 18-months
  Concentration of PTH (pg/ml)
25(OH)D | Baseline, 3, 9 and 18-months
  Concentration of 25(OH)D (ng/mL)
P1NP | Baseline, 3, 9 and 18-months
  Concentration of Procollagen I Intact N-Terminal or P1NP (ug/L )
CTX | Baseline, 3, 9 and 18-months
  Concentration of C-terminal telopeptide or CTX (pg/mL)
TRAP 5b | Baseline, 3, 9 and 18-months
  Concentration of Tartrate-resistant acid phosphatase 5b or TRAP 5bC-Terminal to Intact (U/L)
BSAP | Baseline, 3, 9 and 18-months
  Concentration of Bone-specific alkaline phosphatase or BSAP (mcg/L)
cFGF23 | Baseline, 3, 9 and 18-months
  Concentration of Fibroblast Growth Factor 23 or cFGF23 (pmol/L) and iFGF23 (pg/mL)
Klotho | Baseline, 3, 9 and 18-months
  Concentration of Klotho (pg/mL) and soluble α-Klotho (pg/mL)
Sclerostin | Baseline, 3, 9 and 18-months
  Concentration of Sclerostin and Bioactive Sclerostin (pmol/L)
DKK1 | Baseline, 3, 9 and 18-months
  Concentration of DKK1 (pmol/L)
Fetuin A | Baseline, 3, 9 and 18-months
  Concentration of Fetuin A (ng/mL)
Zinc | Baseline, 3, 9 and 18-months
  Concentration of Zinc (μmol/L)
Irisin | Baseline, 3, 9 and 18-months
  Concentration of Irisin
Serum Calcification Propensity T50 test | Baseline, 3, 9 and 18-months
  Serum Calcification Propensity T50 test (minutes)
Hemoglobin (Hb) | Baseline, 3, 9 and 18-months
  Concentration of Hemoglobin (g/dl)
Hematocrit (Ht) | Baseline, 3, 9 and 18-months
  Concentration of Hematocrit (%)
Plates (PLTS) | Baseline, 3, 9 and 18-months
  Concentration of plates (g/L)
Reticulocytes | Baseline, 3, 9 and 18-months
  Concentration of reticulocytes (%)
Iron | Baseline, 3, 9 and 18-months
  Concentration of iron (µg/dL)
Ferritin | Baseline, 3, 9 and 18-months
  Concentration of ferritin (ng/ml )
Transferrin | Baseline, 3, 9 and 18-months
  Concentration of transferrin (mg/dL)
Transferrin Saturation | Baseline, 3, 9 and 18-months
  Transferrin saturation (%)
Albumin | Baseline, 3, 9 and 18-months
  Concentration of Albumin (g/dl)
KT/V | Baseline, 3, 9 and 18-months
  Level of KT/V
Aluminium | Baseline, 3, 9 and 18-months
  Concentration of aluminium (mcg/L)
C-reactive Protein (CRP) | Baseline, 3, 9 and 18-months
  Concentration of C-reactive Protein (mg/L)
Cholesterol | Baseline, 3, 9 and 18-months
  Concentration of cholesterol (mg/dl)
Triglycerides | Baseline, 3, 9 and 18-months
  Concentration of triglycerides (mg/dl)
Cholesterol HDL | Baseline, 3, 9 and 18-months
  Concentration of Cholesterol HDL (mg/dl)
Cholesterol LDL | Baseline, 3, 9 and 18-months
  Concentration of Cholesterol LDL (mg/dl)
Vascular Calcification | Baseline, 18-months
  Number of participants with vascular calcification (Aorta and Iliac arteries) by lateral Dorsal Lumbar spine x-Ray.
Vertebral Fractures | Baseline, 18-months
  Changes from baseline prevalence Vertebral Fractures (VFs, quantitative vertebral morphometry using dedicated software) by lateral Dorsal Lumbar spine x-Ray
BMD: Bone Mineral Density | Baseline, 18-months
  Changes from baseline Total Hip, Femoral neck Bone Mass Density (BMD) by Dual-energy X-ray absorptiometry (DEXA) including Trabecular Bone Score where it will be available (TBS).
Association between Verterbal Fractures and Vascular Calcificatiom | Baseline, 18-months
  To evaluate the relationship of bone vascular biomarkers on clinical outcomes: VFs and VCs
Novel quantitative computer-assisted scoring method for vascular calcifications. | Baseline, 18-months
  To compare a novel quantitative computer-assisted scoring method for vascular calcifications with a three-dimensional assessment from CT data
Effect of Etelcalcetide on cardiovascular events and all-cause mortality. | Baseline, 18-months
  Effect of Etelcalcetide on the number of cardiovascular events and on the number of all-cause deaths.
Etelcalcetide Safety: Number of participants with treatment-related adverse events. | Baseline, 18-months
  The outcome can identify potential adverse events, such as: Blood calcium decrease, Muscle spasms, Diarrhea, Nausea, Vomiting, Headache, Hypocalcaemia, Hypertension, Hypotension, Arteriovenous fistula site complication, Pain in extremity, Paresthesia, Back pain, Upper respiratory tract infection.